CLINICAL TRIAL: NCT03281577
Title: A Dose-Ranging, Randomized, Parallel, Placebo-Controlled Study to Assess the Effect of TAK-954 on Gastrointestinal and Colonic Transit in Patients With Diabetic or Idiopathic Gastroparesis
Brief Title: Effect of TAK-954 on Gastrointestinal and Colonic Transit in Diabetic or Idiopathic Gastroparesis Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-954-2003; U1111-1200-9396 (Registry Identifier: WHO)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Gastroparesis; Idiopathic Gastroparesis
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): TAK-954 placebo-matching, 60-minute infusion, intravenously (IV), once daily on Days 1 to 3.
  Interventions: Drug: Placebo
- TAK-954 0.1 mg (Experimental): TAK-954 0.1 mg, 60-minute infusion, IV, once daily on Days 1 to 3.
  Interventions: Drug: TAK-954
- TAK-954 0.3 mg (Experimental): TAK-954 1 mg, 60-minute infusion, IV, once daily for up to 3 days.
  Interventions: Drug: TAK-954
- TAK-954 1 mg (Experimental): TAK-954 1 mg, 60-minute infusion, IV, once daily on Days 1 to 3.
  Interventions: Drug: TAK-954

INTERVENTIONS:
Drug: TAK-954 — TAK-954 IV infusion.
  Arms: TAK-954 0.1 mg; TAK-954 0.3 mg; TAK-954 1 mg
Drug: Placebo — TAK-954 placebo-matching IV infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the dose-dependent effects of TAK-954 on gastric emptying time of solids in participants with diabetic or idiopathic gastroparesis assessed by scintigraphy.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-954. TAK-954 is a serotonin (5 HT4) receptor agonist and is being tested to treat people who have diabetic or idiopathic gastroparesis and who previously reported delay in stomach emptying. This study will look at the gastric emptying time of solids in people who take TAK-954 or placebo.

The study will enroll approximately 41 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-954 0.1 mg
* TAK-954 0.3 mg
* TAK-954 1 mg
* Placebo (dummy inactive solution) - this is a solution that looks like the study drug but has no active ingredient.

This single center trial will be conducted in the United States. The duration of treatment is 3 days and the overall period of evaluation is up to 28 days. The participants will be contacted by telephone (Days 10 to 14) for follow-up assessment. There will be another follow-up phone call for women of childbearing potential (Days 38 to 43).

ELIGIBILITY:
Inclusion Criteria:

1. Has diabetes mellitus with symptoms of gastroparesis and previously documented gastric emptying delay or previously documented idiopathic gastroparesis in the last 5 years.
2. Has a body mass index (BMI) greater than or equal to (>=) 16 and less than or equal to (<=) 40 kilogram per square meter (kg/m^2) at the Screening Visit.

Exclusion Criteria:

1. Has glycosylated hemoglobin (HbA1c) greater than (>) 12 percent (%).
2. Has other structural diseases/conditions that affect the gastrointestinal (GI) system.
3. Are unable to withdraw drugs known to alter GI transit 48 hours prior to the study.
4. Has clinically significant abnormal baseline safety laboratory values.
5. Has preexisting hepatic disease that meets Child-Pugh Class B (moderate; total score 7 to 9 points) or C (severe; total score 10 to 15 points).
6. Are without known preexisting hepatic disease who have 1 or more of the following:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 times the upper limit of normal (ULN).
   * Bilirubin >1.5 times the ULN unless due to Gilbert's syndrome.
   * International normalized ratio (INR) >1.5 unless on anticoagulation therapy.
7. Has QT intervals with Fridericia correction method (QTcF) interval (>=) 460 millisecond (msec) or with other factors that increase the risk of QT prolongation or arrhythmic events at screening. Note: Participants with bundle branch block and a prolonged QTc interval, or with QTcF between 450 and 460 msec, should be reviewed by the Medical Monitor for potential inclusion.
8. Has second or third degree atrioventricular (AV) block; AV disassociation; >5 beats of non-sustained VT at a rate >120 beats per minute (bpm); Electrocardiogram (ECG) changes consistent with acute myocardial ischemia or infarction.
9. Has cardiac history that includes conditions requiring heart rate control (example, atrial fibrillation, atrial flutter, ventricular tachycardia, or other tachyarrhythmias).
10. Has clinical evidence (including physical examination, ECG, clinical laboratory value and review of the medical history) of significant cardiovascular, respiratory, moderate or severe renal insufficiency (creatinine clearance <=60 mL/min), hematological, neurological, or psychiatric disease, or other disease that interferes with the objectives of the study.
11. If female, are pregnant or lactating or intending to become pregnant before participating in this study, during the study, and 4 to 5 days (5 half-lives) PLUS 30 days after last dose of the study drug; or intending to donate ova during such time period.
12. Are considered by the investigator to be alcoholics not in remission or known substance abusers. Have a history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to: beer [354 milliliter per [mL/] 12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce] per day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Chedid V, Brandler J, Arndt K, Vijayvargiya P, Wang XJ, Burton D, Harmsen WS, Siegelman J, Chen C, Chen Y, Almansa C, Dukes G, Camilleri M. Randomised study: effects of the 5-HT4 receptor agonist felcisetrag vs placebo on gut transit in patients with gastroparesis. Aliment Pharmacol Ther. 2021 May;53(9):1010-1020. doi: 10.1111/apt.16304. Epub 2021 Mar 12. PMID 33711180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 02 January 2018 to 12 July 2019.
Pre-assignment Details: Participants with a diagnosis of diabetic or idiopathic gastroparesis were enrolled and randomized in 1:1:1:1 ratio to receive TAK-954 0.1 mg, 0.3 mg, 1 mg or placebo.
Groups:
- TAK-954 0.3 mg: TAK-954 0.3 mg, 60-minute infusion, IV, once daily on Days 1 to 3.
Period: Overall Study
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Started | 10 | 10 | 9 | 7
Completed | 9 | 10 | 9 | 6
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects who receive at least 1 dose of study drug.
Groups:
- Placebo: TAK-954 placebo-matching, 60-minute infusion, IV, once daily on Days 1 to 3.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg | Total
Number analyzed (Participants) | 10 | 10 | 9 | 7 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (15.67) | 46.8 (12.45) | 42.3 (11.82) | 40.3 (8.75) | 44.3 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 7 | 5 | 30
  Male | 2 | 0 | 2 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 9 | 7 | 34
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 10 | 9 | 7 | 36
Disease History [Count of Participants; unit: Participants] — Participants were categorized based on whether they have idiopathic gastroparesis or diabetic gastroparesis.
  Participants
    Idiopathic Gastroparesis | 7 | 7 | 3 | 5 | 22
    Diabetic Gastroparesis | 3 | 3 | 6 | 2 | 14
Weight [Mean (Standard Deviation); unit: kg] | 68.3 (15.05) | 73.4 (14.57) | 76.5 (17.97) | 62.5 (9.22) | 70.6 (15.07)
Height [Mean (Standard Deviation); unit: cm] | 166.2 (9.37) | 160.7 (7.27) | 165.7 (5.92) | 166.3 (7.57) | 164.6 (7.74)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight (kg)/height (m)^2
  kg/m^2 | 24.8 (4.88) | 28.4 (5.50) | 27.7 (5.44) | 22.6 (3.15) | 26.1 (5.24)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Half-emptying Time (T1/2) of Gastric Solids
Description: Half-emptying time (t1/2) of gastric solids is the time for half of the ingested solids or liquids to leave the stomach. Scintigraphy assessments were used to evaluate the gastric emptying of solids following a radio-labelled meal. A negative percent change from baseline indicated improvement.
Time Frame: Predose and at multiple time-points post-dose (up to 9 hours) on Day 2
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug. Overall number of participants analyzed is number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 9 | 10 | 9 | 6
percent change | 3.5 (23.71) | -19.8 (14.43) | -25.4 (20.90) | -25.7 (23.56)
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.1 mg; Test type: Superiority; p = 0.0012, ANCOVA — Dunnett's test was used to compare each treatment arm to placebo. Multiplicity Adjusted p-value and 95% confidence interval (CI) are presented; Least Squares Mean Differences = -25.81, 95% CI 2-sided [-41.757 to -9.858] — Linear mixed effects model used for analyses using gastroparesis type [diabetic or idiopathic], age, gender, BMI, baseline as covariate
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.3 mg; Test type: Superiority; p = 0.0018, ANCOVA — Dunnett's test was used to compare each treatment arm to placebo. Multiplicity Adjusted p-value and 95% CI are presented; Least Squares Mean Differences = -27.52, 95% CI 2-sided [-45.224 to -9.813] — Linear mixed effects model used for analyses using gastroparesis type [diabetic or idiopathic], age, gender, BMI, baseline as a covariate
Statistical Analysis 3: Comparison: Placebo vs TAK-954 1 mg; Test type: Superiority; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = -41.76, 95% CI 2-sided [-59.616 to -23.902] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Colonic Geometric Center
Description: The scintigraphic method was used to measure colonic geometric center following a radio-labelled meal. The geometric center (GC) was the weighted average of counts in the different colonic regions, where 0= no radioactivity in the colon and if radioactivity was detected in the colon, 1=all isotope was in the ascending colon and 5=all isotope was in the stool; a high GC indicated faster colonic transit.
Time Frame: 4, 24, and 48 hours post-radiolabeled meal on Day 2
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 10 | 10 | 9 | 7
score on a scale
  Colonic Transit at 4 Hours, Day 2: number analyzed (Participants) | 9 | 10 | 9 | 6
  Colonic Transit at 4 Hours, Day 2 | 0.539 (0.6809) | 1.190 (0.9083) | 1.737 (1.0302) | 1.148 (0.4138)
  Colonic Transit at 24 Hours, Day 2: number analyzed (Participants) | 8 | 10 | 9 | 6
  Colonic Transit at 24 Hours, Day 2 | 1.965 (1.2964) | 3.792 (1.1441) | 3.468 (1.3252) | 2.978 (1.1382)
  Colonic Transit at 48 Hours, Day 2: number analyzed (Participants) | 9 | 10 | 9 | 6
  Colonic Transit at 48 Hours, Day 2 | 3.323 (1.2948) | 4.406 (1.1169) | 4.550 (0.9004) | 3.792 (1.0382)
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.1 mg; Colonic Transit at 4 Hours, Day 2; Test type: Superiority; p = 0.2590, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 0.72, 95% CI 2-sided [-0.364 to 1.795] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.3 mg; Colonic Transit at 4 Hours, Day 2; Test type: Superiority; p = 0.0280, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 1.27, 95% CI 2-sided [0.119 to 2.418] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-954 1 mg; Colonic Transit at 4 Hours, Day 2; Test type: Superiority; p = 0.6882, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 0.45, 95% CI 2-sided [-0.757 to 1.660] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Placebo vs TAK-954 0.1 mg; Colonic Transit at 24 Hours, Day 2; Test type: Superiority; p = 0.0062, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 1.87, 95% CI 2-sided [0.493 to 3.250] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Placebo vs TAK-954 0.3 mg; Colonic Transit at 24 Hours, Day 2; Test type: Superiority; p = 0.1490, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 1.19, 95% CI 2-sided [-0.327 to 2.717] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Placebo vs TAK-954 1 mg; Colonic Transit at 24 Hours, Day 2; Test type: Superiority; p = 0.6285, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 0.63, 95% CI 2-sided [-0.931 to 2.200] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Placebo vs TAK-954 0.1 mg; Colonic Transit at 48 Hours, Day 2; Test type: Superiority; p = 0.0358, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 1.29, 95% CI 2-sided [0.073 to 2.501] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Placebo vs TAK-954 0.3 mg; Colonic Transit at 48 Hours, Day 2; Test type: Superiority; p = 0.0430, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 1.33, 95% CI 2-sided [0.035 to 2.621] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Placebo vs TAK-954 1 mg; Colonic Transit at 48 Hours, Day 2; Test type: Superiority; p = 0.9419, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 0.25, 95% CI 2-sided [-1.107 to 1.611] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Colonic Filling at Hour 6
Description: Colonic filling was estimated as percentage of the radio-labelled meal that reached the colon at Hour 6.
Time Frame: 6 hours post-radiolabel meal on Day 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of radio-labelled food
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 9 | 10 | 9 | 6
percentage of radio-labelled food | 31.3 (25.38) | 55.6 (31.31) | 86.4 (19.76) | 75.3 (31.70)
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.1 mg; Test type: Superiority; p = 0.0436, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 33.12, 95% CI 2-sided [0.799 to 65.439] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.3 mg; Test type: Superiority; p = 0.0007, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 57.98, 95% CI 2-sided [23.555 to 92.396] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-954 1 mg; Test type: Superiority; p = 0.0134, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = 44.44, 95% CI 2-sided [8.249 to 80.629] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Half-emptying Time (T1/2) of Ascending Colon
Description: T1/2 of ascending colon emptying was estimated by analysis of proportionate emptying over time of counts from the colon. Scintigraphy assessments were used to evaluate the emptying of solids or liquids from ascending colon following a radio-labelled meal.
Time Frame: Predose and at multiple time-points post-dose (up to 25 hours) on Days 1, 2 and 3
Population: Full analysis set included all randomized participants who received at least 1 dose of study drug. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Median (Full Range); unit: hours
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 9 | 10 | 9 | 6
hours | 19.1 [2.6 to 36.0] | 5.4 [1.9 to 28.8] | 6.3 [0.6 to 11.0] | 7.4 [0.9 to 13.6]
Statistical Analysis 1: Comparison: Placebo vs TAK-954 0.1 mg; Test type: Superiority; p = 0.0789, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = -10.27, 95% CI 2-sided [-21.507 to 0.960] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-954 0.3 mg; Test type: Superiority; p = 0.0270, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = -13.28, 95% CI 2-sided [-25.242 to -1.314] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-954 1 mg; Test type: Superiority; p = 0.0750, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Least Squares Mean Differences = -11.63, 95% CI 2-sided [-24.206 to 0.952] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: AUCtau: Area Under the Plasma Concentration-Time Curve From Time 0 to t for TAK-954
Time Frame: Predose and at multiple time-points post-dose (up to 25 hours) on Days 1, 2 and 3
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug and had sufficient blood sampling to allow for PK evaluation. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 10 | 9 | 7
h*ng/mL
  Day 1: number analyzed (Participants) | 10 | 8 | 6
  Day 1 | 8.99 (2.110) | 25.79 (8.340) | 83.75 (25.453)
  Day 2: number analyzed (Participants) | 8 | 8 | 5
  Day 2 | 12.16 (3.033) | 33.94 (9.249) | 109.86 (31.009)
  Day 3: number analyzed (Participants) | 9 | 8 | 5
  Day 3 | 15.72 (3.387) | 39.34 (12.699) | 125.88 (34.586)

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-954
Time Frame: Predose and at multiple time-points post-dose (up to 25 hours) on Days 1, 2 and 3
Population: PK analysis set included all participants who received at least 1 dose of study drug and had sufficient blood sampling to allow for PK evaluation. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 10 | 9 | 7
ng/mL
  Day 1: number analyzed (Participants) | 10 | 8 | 7
  Day 1 | 1.637 (0.3918) | 5.346 (1.5797) | 16.029 (2.9239)
  Day 2: number analyzed (Participants) | 9 | 8 | 6
  Day 2 | 1.687 (0.4227) | 5.821 (1.9447) | 15.517 (3.7070)
  Day 3: number analyzed (Participants) | 10 | 8 | 5
  Day 3 | 1.705 (0.3297) | 5.056 (1.5430) | 17.700 (7.1544)

7. Secondary Outcome: Ctrough: Observed Plasma Concentration at the End of a Dosing Interval
Time Frame: At multiple time-points post-dose, up to 9 hours on Day 2 and up to 25 hours on Day 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
Number analyzed (Participants) | 10 | 9 | 7
ng/mL
  Day 2: number analyzed (Participants) | 10 | 9 | 6
  Day 2 | 0.1969 (0.05406) | 0.4364 (0.20371) | 1.6817 (0.47072)
  Day 3: number analyzed (Participants) | 9 | 9 | 5
  Day 3 | 0.2854 (0.10319) | 0.6392 (0.26371) | 2.2620 (0.40493)

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose (Up to 46 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TAK-954 0.1 mg | TAK-954 0.3 mg | TAK-954 1 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/9 | 1/7
Other Adverse Events (participants affected / at risk) | 6/10 | 5/10 | 6/9 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | TAK-954 0.1 mg (N=10) | TAK-954 0.3 mg (N=9) | TAK-954 1 mg (N=7)
Pancreatic enzymes increased (Investigations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | TAK-954 0.1 mg (N=10) | TAK-954 0.3 mg (N=9) | TAK-954 1 mg (N=7)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 4 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 3 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03281577/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT03281577/SAP_001.pdf